CLINICAL TRIAL: NCT02344524
Title: Drainage of Traumatic Hemothorax and Pneumothorax: Small Bore Versus Large Bore Chest Drain- a Randomized Controlled Trial
Brief Title: Drainage of Traumatic Hemothorax and Pneumothorax: Small Bore Versus Large Bore Chest Drain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delhi University (Other)
Responsible Party: Principal Investigator, Sunil Kumar, Director Professor & Head, Department of Surgery, Delhi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRI/2014/07/004795
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Traumatic Hemothorax and Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Small bore chest drain (Experimental): Intercostal drainage for traumatic hemothorax and pneumothorax using small bore chest drain
  Interventions: Device: Intercostal drainage
- Large bore chest drain (Active Comparator): Intercostal drainage for traumatic hemothorax and pneumothorax using large bore chest drain
  Interventions: Device: Intercostal drainage

INTERVENTIONS:
Device: Intercostal drainage — Small bore chest drains are inserted by modified Seldinger's technique. Large bore chest drains are inserted by blunt dissection technique.

SUMMARY:
The purpose of this trial is to study the role of small bore chest drains in draining traumatic hemothorax and pneumothorax.

DETAILED DESCRIPTION:
The precise role of small bore chest drains in treating post traumatic pleural collections, especially hemothorax is not well established. This trial is conducted to study the efficacy and safety profile of small bore chest drains in trauma patients with hemothorax and pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic hemothorax, pneumothorax and hemopneumothorax

Exclusion Criteria:

* Patients with tension pneumothorax
* Patients requiring emergency thoracotomy
* Patients who had undergone chest drain insertion elsewhere
* Patients lost to follow up

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Success rate | 7 days (plus or minus 5 days)
  Complete drainage of traumatic hemothorax and pneumothorax

SECONDARY OUTCOMES:
Procedure time | At the time of the intervention
  Time taken for inserting the chest drain
Iatrogenic injuries | At the time of the intervention
  Insertion related complications
Resolution time | 7 days (plus or minus 5 days)
  Time taken for complete drainage of traumatic hemothorax and pneumothorax
Wound healing time | 10 days (plus or minus 5 days)
  Time taken for the chest drain site wound to heal
Catheter sepsis | 7 days (plus or minus 5 days)
  Identification of infective organisms from catheter tip based on culture following chest drain removal

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Kumar, MS, Principal Investigator — Delhi University
Locations (1):
- University College of Medical Sciences & GTB Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Yi JH, Liu HB, Zhang M, Wu JS, Yang JX, Chen JM, Xu SX, Wang JA. Management of traumatic hemothorax by closed thoracic drainage using a central venous catheter. J Zhejiang Univ Sci B. 2012 Jan;13(1):43-8. doi: 10.1631/jzus.B1100161. PMID 22205619